CLINICAL TRIAL: NCT07200739
Title: Development and Validation of Non-Invasive Danish Language and Speech Biomarkers for Neurodegenerative Disease Classification by Means of Automatic Speech Recognition With Artificial Intelligence (DetectAI)
Brief Title: Speech-Based Artificial Intelligence for Detection of Dementia in Danish Patients
Acronym: DetectAI
Status: Enrolling by invitation | Type: Observational
Sponsor: Zealand University Hospital (Other)
Collaborators: DemensAI ApS (private tech partner, Denmark) (Unknown)
Responsible Party: Sponsor
Other Study IDs: SJ-1107
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Dementia (Diagnosis); Alzheimer Dementia (AD); Vascular Dementia (VaD); Lewy Body Dementia (LBD); Frontotemporal Dementia (FTD); Mild Cognitive Impairment (MCI); Depression - Major Depressive Disorder
Keywords: artificial intelligence; speech-based artificial intelligence; artificial intelligence in dementia diagnostics; artificial intelligence for dementia screening; artificial intelligence for dementia classification; speech based artificial intelligence; dementia; Vascular dementia (VaD); Alzheimer dementia (AD); Lewy Body Dementia (LBD); Frontotemporal Dementia (FTD); Mild Cognitive Impairment (MCI); Depression - Major Depressive disorder; Dementia (diagnosis)
MeSH Terms: conditions — Dementia; Disease; Alzheimer Disease; Dementia, Vascular; Lewy Body Disease; Frontotemporal Dementia; Cognitive Dysfunction | interventions — Blood Specimen Collection; Diploidy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy Controls: n~40
  Interventions: Diagnostic Test: Mini-mental State Examination; Diagnostic Test: Addenbrooke's Cognitive Examination; Other: Speech task - Picture Description; Other: Speech task - Story Retellling; Diagnostic Test: MRI; Diagnostic Test: blood sampling; Diagnostic Test: Depression screening; Other: Somatic- and neurological examination
- New Referrals: New Referrals to the memory clinic. Diagnosis unknown at the time of enrollment. N~200
  Interventions: Diagnostic Test: Mini-mental State Examination; Diagnostic Test: Addenbrooke's Cognitive Examination; Other: Speech task - Picture Description; Other: Speech task - Story Retellling
- Participants from follow-up: Participants with a clinical consensus diagnosis of either Alzheimer's dementia, Vascular dementia, Lewy body Dementia, Frontotemporal Dementia, Mild Cognitive Impairment or Depression. Diagnosis must be established in the memory clinic at ZUH within the past 6 months at the time of enrollment. N~100
  Interventions: Diagnostic Test: Mini-mental State Examination; Other: Speech task - Picture Description; Other: Speech task - Story Retellling; Other: Fluency tasks

INTERVENTIONS:
Diagnostic Test: Mini-mental State Examination — Participants will be recorded during the test in order til allow the AI to learn and analyze speech patterns.
  Other Names: MMSE
Diagnostic Test: Addenbrooke's Cognitive Examination — Participants will be recorded during the test in order til allow the AI to learn and analyze speech patterns.
  Other Names: ACE
  Groups: Healthy Controls; New Referrals
Other: Speech task - Picture Description — Participants will be asked to describe the Cookie Theft Picture from the Boston Diagnostic Aphasia Examination. The task will take 2 minutes. Participants will be recorded during the speech task in order to allow the AI to learn and analyze the speech patterns.
Other: Speech task - Story Retellling — Participants will be asked to retell the fairy-tale "Cinderella", based on pictures that summarize the fairy-tale. In case "Cinderella" is not known, participants are asked to tell a story with a start, a middle and an end based on the provided pictures. The task will take 4 minutes. Participants will be recorded during the speech task in order to allow the AI to learn and analyze the speech patterns.
Other: Fluency tasks — Two fluency tasks from the Addenbrooke's Cognitive Examination. First, the participant is asked to name as many animals as possible within 1 minutes. Next the participant is asked to name as many words starting with "S" as possible within 1 minute.
  Participants will be recorded during the tasks in order to allow the AI to learn and analyze speech patterns.
  Groups: Participants from follow-up
Diagnostic Test: MRI — For healthy controls an MRI will be conducted to provide comparable imaging and as part of screening to ensure they do not meet exclusion criteria (neuroradiological findings that could affect cognitive functions).
  For participants in the follow-up or new referral cohorts, imaging will be performed as part of the standard diagnostic battery and results will be obtained from the electronic journal.
  Groups: Healthy Controls
Diagnostic Test: blood sampling — Healthy control participants will undergo a standard blood test panel commonly used in dementia diagnostics. The panel includes complete blood counts, inflammatory markers, kidney- and liver function markers, thyroid-stimulating hormone (TSH), vitamine B12 and folate. These tests are performed to exclude underlying medical conditions that could mimic cognitive impairment.
  For participants in the follow-up or new referral cohorts, blood sampling will be performed as part of the standard diagnostic battery and results will be obtained from the electronic journal.
  Groups: Healthy Controls
Diagnostic Test: Depression screening — Performed on healthy controls to rule out depression using either the geriatric depression scale (GDS) for patients > 65 year of age or the Major Depression Index (MDI) for patiens <65 year of age.
  For participants in the follow-up or new referral cohorts, depression screening will be performed as part of the standard diagnostic battery and results will be obtained from the electronic journal.
  Groups: Healthy Controls
Other: Somatic- and neurological examination — Healthy controls will undergo a standard somatic and neurological examination to exclude conditions that may affect cognition. This includes basic neurological assessment and clinical evaluation of general health status.
  For participants in the follow-up or new referral cohorts, a somatic and neurological examination will be performed as part of the standard diagnostic battery and results will be obtained from the electronic journal
  Groups: Healthy Controls

SUMMARY:
The goal of this observational study is to develop and test an artificial intelligence (AI) model that can detect signs of dementia and related conditions from speech recordings. The main question is whether a speech-based AI model can correctly tell apart people with normal memory and thinking from those with cognitive impairment.

The study will also explore whether the AI can distinguish dementia from depression, separate different dementia subtypes, and identify which people with Mild Cognitive Impairment (MCI) are likely to develop dementia.

Participants will complete short memory and speech tasks while being recorded. The AI model will analyze these recordings to learn patterns linked to different diagnoses. At the end of the study, its accuracy will be tested on new participants.

DETAILED DESCRIPTION:
Background Dementia is a growing public health challenge, and early and accurate diagnosis is essential for effective care and potential future disease-modifying treatments. Current diagnostic pathways are resource-intensive and associated with long waiting times. Speech reflects cognitive functioning, and recent international studies have shown that AI can detect dementia-related patterns in speech recordings with promising accuracy. This study aims to develop and validate a speech-based AI model in a Danish setting, providing a non-invasive and scalable screening tool for use in primary care.

Phases one This protocol describes the first phase of our study which is expected to be completed in two separate phases.

In phase one we seek to train an AI model to analyse speech data from participants with cognitive impairment and compare it to speech data from healthy control participants, as is detailed through this protocol. If the method is validated, we will continue to phase two.

Future work In phase two we expect to conduct an external validation. The AI model analysis will be performed on 200 participants in the primary care sector referred for dementia evaluation. The results of the AI analysis will be compared against the final gold standard consensus diagnosis.

Phase two will have a separate protocol which will be worked up based on the results from phase one.

Elaboration of time perspective Other: Hybrid design. Most participants will be included in a cross-sectional case-control study (single speech recording). For participants with MCI, follow-up data will be collected within the study period to assess progression to dementia, allowing evaluation of the model's ability to distinguish progressive from non-progressive MCI.

ELIGIBILITY:
Inclusion Criteria:

* Age > 50 years
* Fluent in Danish
* Minimum 7 years of schooling

For participants from the follow-up cohort:

* A consensus diagnosis of either AD, VaD, LBD, FTD, MCI or depression established at the memory clinic within 6 months prior to enrollment

For participants from the healthy control cohort:

* No known cognitive impairment or affective disorder

Exclusion Criteria:

* Significantly impaired vision or hearing (to the extent that the participant cannot participate in the linguistic AI analysis)
* Participants unable to give consent

Participants from follow-up and new referrals cohort:

* MMSE score < 16
* Participants with multiple diagnoses (eg. mixed dementia or AD with concurrent depression)

For participants from the new referrals cohort:

* Participants falling outside of the six categories included in the study (AD, VaD, LBD, FTD, MCI, Depression)
* Participants where it is obvious at baseline that they will not fall within the above categories (can be excluded before clinical consensus diagnosis is given)

For participants from the healthy control cohort:

* MMSE <26 and ACE <90
* GDS score indicating depression (6 or higher)
* Clinical, laboratory or neuroradiological findings that could affect cognitive functions

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants are recruited from patients who are followed at- or referred to the memory clinic at Zealand University Hospital. Age and gender matched healthy controls are recruited from the participants' relatives.
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Accuracy of AI model in classifying cognitive impairment vs. unimpaired cognition | At baseline (speech recording)
  Measured by sensitivity, specificity, AUR-ROC of AI predictions compared to clinical consensus diagnosis, using baseline speech recordings from participants.
  Model performance will be measured after database lock at study completion.

SECONDARY OUTCOMES:
Accuracy for dementia vs. depression | At baseline (speech recording)
  Measured by sensitivity, specificity, AUR-ROC of AI predictions compared to clinical consensus diagnosis, using baseline speech recordings from participants. Model performance will be measured after database lock at study completion.
Sub-classification of Mild Cognitive Impairment (MCI) into progressive vs. non-progressive | At baseline (speech recording) and up to 12 months after enrollment (to determine progression)
  Measured by sensitivity, specificity, AUR-ROC of AI predictions compared to clinical consensus diagnosis, using baseline speech recordings from participants. Model performance will be measured after database lock at study completion.
  Progression is defined as new dementia diagnosis during study period.
Classification of dementia subtypes (AD, VaD, LBD, FTD) | At baseline (speech recording)
  Measured by sensitivity, specificity, AUR-ROC of AI predictions compared to clinical consensus diagnosis, using baseline speech recordings from participants. Model performance will be measured after database lock at study completion.
Comparison with established biomarkers | At baseline, or at time of biomarker testing if performed after baseline
  Differences in diagnostic accuracy between AI predictions and state-of-the-art biomarkers for dementia diagnosis
Feature importance analysis | At baseline (speech recording)
  Feature importance will be evaluated using interpretability analyses (e.g. permutation importance, SHAP values, and/or ablation of feature groups) to quantify the contribution of acoustic and linguistic features to the model's predictions.

OTHER OUTCOMES:
Contribution of individual speech tasks to AI model performance | At baseline (speech recording)
  Contribution of individual speech tasks will be evaluated by comparing model performance (e.g. accuracy, sensitivity, specificity, AUC-ROC) when trained and tested on subsets of speech tasks (memory tests, story recall, picture description). This will identify which tasks provide the strongest diagnostic signal.
Number of tasks required for optimal accuracy | At baseline (speech recording)
  Evaluation of whether a reduced set of speech tasks provide accuracy comparable to the full test battery.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Høgh, MD, PhD, Assoc Prof, Principal Investigator — Zealand University Hospital
Locations (1):
- Zealand University Hospital, Roskilde, Region Sjælland, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dargaud L, Partal A, Birn A, & Detlefsen S. N. (2023). Developing a Spontaneous Speech-based Artificial Intelligence for Alzheimer's Disease Detection. Transatlantic Telehealth Research Network (TTRN) International Scientific Conference 2023, Journal of the International Society for Telemedicine and eHealth.
- [Background] Lanzi AM, Saylor AK, Fromm D, Liu H, MacWhinney B, Cohen ML. DementiaBank: Theoretical Rationale, Protocol, and Illustrative Analyses. Am J Speech Lang Pathol. 2023 Mar 9;32(2):426-438. doi: 10.1044/2022_AJSLP-22-00281. Epub 2023 Feb 15. PMID 36791255
- [Background] Li J, Song K, Zheng B, Li D, Wu X, Meng H. Leveraging Pretrained Representations with Task-related Keywords for Alzheimer's Disease Detection. arXiv preprint. 2023.
- [Background] Luz S, Haider F, de la Fuente Garcia S, Fromm D, MacWhinney B. Detecting cognitive decline using speech only: The ADReSSo challenge. arXiv preprint 2021.
- [Background] Luz S, Haider F, Fromm D, Lazarou I, Kompatsiaris I, Macwhinney B. An Overview of the ADReSS-M Signal Processing Grand Challenge on Multilingual Alzheimer's Dementia Recognition Through Spontaneous Speech. IEEE Open J Signal Process. 2024;5:738-749. doi: 10.1109/ojsp.2024.3378595. Epub 2024 Mar 18. PMID 38957540
- [Background] Bex T. Comprehensive Guide to Multiclass Classification With Sklearn. Towards Data Science. 2021.
- [Background] Nicholas LE, Brookshire RH. A system for quantifying the informativeness and efficiency of the connected speech of adults with aphasia. J Speech Hear Res. 1993 Apr;36(2):338-50. doi: 10.1044/jshr.3602.338. PMID 8487525
- [Background] Buderer NM. Statistical methodology: I. Incorporating the prevalence of disease into the sample size calculation for sensitivity and specificity. Acad Emerg Med. 1996 Sep;3(9):895-900. doi: 10.1111/j.1553-2712.1996.tb03538.x. PMID 8870764
- [Background] Chen J, Ye J, Tang F, Zhou J. Automatic Detection of Alzheimer's Disease Using Spontaneous Speech Only. Interspeech. 2021 Aug-Sep;2021:3830-3834. doi: 10.21437/interspeech.2021-2002. PMID 35493062
- [Background] Agbavor F, Liang H. Predicting dementia from spontaneous speech using large language models. PLOS Digit Health. 2022 Dec 22;1(12):e0000168. doi: 10.1371/journal.pdig.0000168. eCollection 2022 Dec. PMID 36812634
- [Background] de la Fuente Garcia S, Ritchie CW, Luz S. Artificial Intelligence, Speech, and Language Processing Approaches to Monitoring Alzheimer's Disease: A Systematic Review. J Alzheimers Dis. 2020;78(4):1547-1574. doi: 10.3233/JAD-200888. PMID 33185605
- See also: Website of collaborator, DemensAI SPs (responsible party for training and testing the AI model) — https://www.demensai.dk/